CLINICAL TRIAL: NCT04041544
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SN1011 Following Single and Multiple Oral Dose Administration
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Health Subject
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SinoMab BioScience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SN1011-101
Record Dates: First submitted 2019-07-23; First posted 2019-08-01 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-07

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: In total there are planned to be 2 parts to the study. Part A will look at the effects of a single dose of the study drug and Part B will look at the effects of multiple doses of the study drug.
Who Masked: Participant, Investigator
Masking Description: In each dose panel in this study, eight healthy subjects will be randomized in a 6:2 ratio to receive XNW3009 or placebo in SAD and MAD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SN1011 (Active Comparator): 5 Cohort for Part A:25mg once a day,50mg once a day, 100mg once a day, 150mg once a day, 200mg once a day 4 Cohort for Part B : 50mg once a day, 100mg once a day, 200mg once a day, 100mg twice a day
  Interventions: Drug: SN1011
- SN1011 placebo (Placebo Comparator): 5 Cohort for Part A:25mg once a day,50mg once a day, 100mg once a day, 150mg once a day, 200mg once a day 4 Cohort for Part B : 50mg once a day, 100mg once a day, 200mg once a day, 100mg twice a day
  Interventions: Drug: SN1011 placebo

INTERVENTIONS:
Drug: SN1011 — SN1011 will be supplied to the Pharmacy as 25 mg and 100 mg capsules.
  Arms: SN1011
Drug: SN1011 placebo — The placebo to be used in this study will be identical to SN1011, minus the active ingredient.
  Arms: SN1011 placebo

SUMMARY:
SN1011 (the study drug), is currently being developed by Sinomab as a new drug for treating autoimmune disease (diseases occurring when your body's natural immune/defence mechanism attacks healthy tissue and nerves), such as rheumatoid arthritis (RA). RA causes recurrent joint pain and swelling, particularly in the hands and feet, and can lead to bone erosion and joint deformity.

SN1011 is known as a BTK inhibitor. Bruton's tyrosine kinase (BTK) is an enzyme that plays a key role in B-cell development, and B-cells play an important role in immunity throughout the body. It is thought that blocking the BTK signal may inhibit disease progression in people with RA and may even resolve the disease.

The purpose of this research study is to assess the safety and tolerability of SN1011 as well as the pharmacokinetics (PK - how your body handles the study drug) and pharmacodynamics (PD - how the study drug affects your body) of the study drug. The investigators are doing this study in healthy men and women.

DETAILED DESCRIPTION:
This study will compare SN1011 with placebo. A placebo has no active drug in it. One group of participants will take SN1011 and another group will take the placebo. The effects seen in participants taking the study drug will be compared to the effects seen in participants who are taking the placebo.

This study will look at how participants react to and how the human body uses SN1011 at different dose levels.

The design of the study is double-blind, randomised and placebo-controlled. In total there are planned to be 2 parts to the study. Part A will look at the effects of a single dose of the study drug and Part B will look at the effects of multiple doses of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Able to give signed written informed consent form
* Body mass index (weight [kg]/height [m]2) within 18.0 to 30.0 kg/m2 (inclusive);
* Blood pressure < 140/90 mmHg at screening and heart rate <100 bpm. One repeat assessment is permitted;
* No clinically significant abnormalities in the 12-lead ECG.
* Creatinine clearance ≥ 90 mL/min at screening;
* Overtly healthy as determined by medical evaluation including medical history and physical examination at screening;
* Have clinical laboratory test results within the study site's normal reference range for: absolute neutrophil count, potassium, liver and kidney function tests. No other screening clinically significant abnormal laboratory tests results. Two repeat assessments are permitted at the discretion of the investigator;
* If male, be willing to remain abstinent
* If female, be of non-childbearing potentia.

Exclusion Criteria:

* History of severe drug or excipient allergy, or hypersensitivity to SN1011 capsules or other BTK inhibitors;
* History of stomach or intestinal surgery or resection
* Current or chronic history of liver disease or known hepatic or biliary abnormalities;
* Current or history of cardiac arrythmias;
* Recent or current serious infection;
* Have had symptomatic herpes zoster infection within 12 weeks of screening;
* Current or history autoimmune disease, or suspected autoimmune disease;
* Presence of cataract(s) or prior history of cataract surgery;
* Recent administration or plans to receive administration of live vaccine;
* Major illness or surgery (except for minor outpatient surgery) within 3 months of study Day 1, or planned surgery during study;
* Intolerance to direct venipuncture;
* Known or suspected history of drug abuse within the past 2 years
* Participation in any clinical study with an investigational drug, biologic or device within 4 weeks;
* Positive screening test for serum hepatitis B surface antigen, hepatitis C antibody or human immunodeficiency virus (HIV);
* Malignancy within 5 years of screening visit (excluding non-melanoma skin cancer that has been resected);
* Evidence of active or latent tuberculosis (TB);
* Pregnant or lactating women;
* Subject who is considered unsuitable for participating in the study in the opinion of investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate incidence and severity of adverse events | From day1 of study drug dosing to day4 for part A.
  An AE is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Evaluate incidence and severity of adverse events | From day1 of study drug dosing to day 13 for part B.
  An AE is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.
Evaluate clinically significant changes from baseline in physical examinations | From day1 of study drug dosing to day4 for part A.
  physical examinations will be performed by a study delegated registered physician.Any findings made during the physical examination must be noted regardless of if they are part of the subject's medical history.
Evaluate clinically significant changes from baseline in physical examinations | From day1 of study drug dosing to day 13 for part B.
  physical examinations will be performed by a study delegated registered physician.Any findings made during the physical examination must be noted regardless of if they are part of the subject's medical history.

SECONDARY OUTCOMES:
Pharmacokinetic Assessments of Maximum plasma concentration (Cmax) | From day1 of study drug dosing to day4 for part A, from day1 of study drug dosing to day 13 for part B.
  To lower the risk of volunteers in this study, exposure of SN1011 will be monitored in the whole study and daily exposure calculated through maximum plasma concentration of SN1011 (Cmax)
Pharmacokinetic Assessments of Time to maximum plasma concentration (tmax) | From day1 of study drug dosing to day4 for part A, from day1 of study drug dosing to day 13 for part B.
  Exposure of SN1011 will be monitored in the whole study and daily exposure calculated through area under the plasma concentration
Pharmacokinetic Assessments of Area under the plasma concentration time curve (AUC) | From day1 of study drug dosing to day4 for part A, from day1 of study drug dosing to day 13 for part B.
  Exposure of SN1011 will be monitored in the whole study and daily exposure calculated through area under the plasma concentration time

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, West Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No